CLINICAL TRIAL: NCT04350294
Title: Children and Adolescents With Parental Mental Illness: Measuring Vocal Brain Development in Babies of Mothers Who Have Experienced Serious Mental Illness
Brief Title: Measuring Development of Brain Responses to Vocal Sounds in Babies of Mums With Mental Illness
Acronym: CAPRI-Voc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Kathryn Abel, Professor, University of Manchester
Other Study IDs: 212715
Record Dates: First submitted 2020-04-06; First posted 2020-04-17 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Mental Disorders, Severe
Keywords: Psychosis; Schizophrenia; Depression; Bipolar; Anxiety; Obsessive Compulsive Disorder
MeSH Terms: conditions — Mental Disorders; Psychotic Disorders; Schizophrenia; Depression; Anxiety Disorders; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Serious Mental Illness *RECRUITMENT IN THIS GROUP IS CLOSED: Mothers with a serious mental illness*
  *received hospitalisation, treatment or intervention from a secondary care (mental health) service in the last 5 years.
- Healthy Controls: Mothers with no history of mental illness, who have given birth since February 2021

SUMMARY:
CAPRI-Voc examines the differences in how speech and environmental sounds are processed in the infant brain as they grow from 9 to 12 months. The main aim of our research is to see whether serious mental illness or other factors influence this development in children. This means we are looking for new mums and their infants who have not experienced mental illness.

DETAILED DESCRIPTION:
A delay in the development of language can make it hard for individuals to socialise and learn. While many children thrive, some children who live with a parent suffering from a mental illness develop difficulties with language and communication. Unfortunately, language delay is often missed until children are at school. By then, treatment options may be more limited and less effective. These children and their families would do better if they had more support early on. There is a lack of research in this area so we are cannot tell whether an individual child is at more risk or whether they have protective qualities. We need to know this to plan treatment and start it early because the earlier the help, the better the results.

Therefore, our study aims to identify children who will be most at risk of difficulties or delays in their language. It will also examine the effects of mental illness and other factors in mothers in the child's language and communication abilities. This will help us to design better treatments for the most at risk children because identifying them when they are infants means we can help their cognitive, development and language skills earlier.

To do this, we use a form of brain imaging called functional Near-Infrared Spectroscopy (fNIRS). It is a safe, non-invasive technique that records brain responses. When nerve cells in our brains are active, the supply of blood increases to those tissues. Our equipment detects these changes in blood flow by shining light onto the scalp. fNIRS has been safely used with thousands of infants worldwide. It is a common tool in neonatal and intensive care units and there are no side effects of fNIRS.

We ask your baby to put a cap on which has light sensors. Whilst baby has the cap on, we get them to watch 2 six-minute videos which have different sounds playing. Here, we will be able to see whether the baby can tell the difference between vocal sounds and environmental sounds (like traffic), as well as the differences in emotional speech (i.e. happy, sad and neutral speech).

As well as measuring baby's brain activity, we also ask mum questions about herself and video a 6-minute play session between mum and baby. Finally, we carry out a play session to measure baby's development. All assessments are done with the utmost care and mum is always present to make sure everyone is comfortable.

ELIGIBILITY:
***If you have given birth in or after February 2021 and are interested in participating, please contact our research team.***

Inclusion Criteria:

* Capacity to consent for themselves and their baby
* Proficiency in English

Exclusion Criteria:

* Women whose baby is permanently removed from their care
* Women with a primary diagnosis of substance/alcohol abuse or dependence in the last year
* Women with a primary diagnosis of anorexia/bulimia nervosa
* Women with a primary diagnosis of a personality disorder, psychological development or somatoform disorders
* Infants with congenital malformations, severe chronic illness, and developmental disorders

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We are interested in recruiting all women who have given birth since February 2021*
  Please contact the our team if you have any questions about your suitability for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
functional near infrared spectroscopy (fNIRS) to assess changes in neural responses over time | When the child is 9 months and 12 months old
  Baby will listen to vocal, non vocal, and emotional speech sounds for around 12 minutes. fNIRS uses near infrared light to capture changes in blood oxygenation in response to the sounds which is analogous to brain function.
  We are only assessing brain responses to the auditory stimuli played, a video is used to keep the baby's attention on the task

SECONDARY OUTCOMES:
Bayley scale of infant and toddler development III | When the child is 12 months old
  A research tool involving standard series of measurements (games/tasks) to assess the cognitive and language development of children. This scale is designed to be used on children up to 3-4 years of age, therefore, the more tasks completed by a child the greater their cognitive or language ability.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Abel, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- See also: CAPRI-Voc website — https://sites.manchester.ac.uk/capri-voc/